CLINICAL TRIAL: NCT05529030
Title: COVID-19 Booster Readiness Survey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Michelle N. Meyer, Faculty Co-Director, Behavioral Insights Team, Geisinger Clinic, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0726
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Vaccination Refusal
Keywords: Communication; Surveys and Questionnaires; Vaccination; Economics, Behavioral
MeSH Terms: conditions — Vaccination Refusal; Communication; Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know that there are different versions of surveys
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard question (No Intervention): Question with no additional text or framing
- Question with salient Omicron message (Experimental): Question indicates that the bivalent booster can protect the respondent from the Omicron variant
  Interventions: Behavioral: Salience of Omicron variant; Behavioral: Self-protection message
- Question with patient protection message (Experimental): Question indicates that the bivalent booster can protect patients (only presented to patient-facing employees)
  Interventions: Behavioral: Other-protection message
- Question with salient Omicron and patient protection message (Experimental): Question indicates that the bivalent booster can protect patients from the Omicron variant (only presented to patient-facing employees)
  Interventions: Behavioral: Salience of Omicron variant

INTERVENTIONS:
Behavioral: Salience of Omicron variant — The message mentions the Omicron variant, which can be a fear appeal or make salient the reason for the new booster
  Arms: Question with salient Omicron and patient protection message; Question with salient Omicron message
Behavioral: Self-protection message — The message makes a reference to protecting one's self
  Arms: Question with salient Omicron message
Behavioral: Other-protection message — The message makes a reference to protecting others (patients)
  Arms: Question with patient protection message

SUMMARY:
The purpose of this administrative survey is to inform health system logistics by assessing the attitudes towards towards the bivalent COVID-19 boosters held by healthcare workers (HCWs) at a large, rural health system. It will also test, prospectively, the effect on interest in the bivalent COVID-19 booster of different framing approaches in a survey question sent to employees of a large, rural health system.

DETAILED DESCRIPTION:
The Food and Drug Administration has authorized two bivalent COVID-19 boosters with the expectation that the Centers for Disease Control will soon recommend them. The researchers plan to survey the HCWs at a large, rural health system on their attitudes on the bivalent booster.

This survey will gather data on HCWs' interest in a bivalent booster, reasons for hesitancy, risk perception about COVID-19 infection and its complications, and prior COVID-19 infection and vaccination.

Respondents will also be randomly assigned to see different versions of the question asking if they are interested in a bivalent booster with different framing approaches, such as protection of the self or protection of patients (for patient-facing employees). Information on prior vaccination and perceptions of risk will also be gathered and used as covariates in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Employee at the health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12036 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Count of employees who indicate interest in the booster | 14 days
  Number of employees who indicate that they plan to get the booster when it is available

CONTACTS AND LOCATIONS:
Overall Officials: Michelle N Meyer, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT05529030/SAP_000.pdf